CLINICAL TRIAL: NCT02074761
Title: Evolusion Study Using the Zyga SImmetry Sacroiliac Joint Fusion System
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Surgalign Spine Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 007-002
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: sacroiliac joint fusion; SIJ fusion; SI joint; SIJ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SImmetry Implant: Subjects who are indicated for the SImmetry device and meet the inclusion/exclusion criteria will receive a SImmetry implant.
  Interventions: Device: SImmetry

INTERVENTIONS:
Device: SImmetry — The SImmetry device is commercially available. The implanted devices consist of a range of threaded, self-tapping, cannulated implants designed to transfix the sacrum and ilium, providing stability for intra-articular fusion.
  The SImmetry Surgical Instruments include standard manual surgical instruments used to access and prepare the sacroiliac joint space for intra-articular fusion.

SUMMARY:
Sacroiliac joint pain reduction and radiographic evidence of SIJ fusion will be collected to evaluate clinical performance of the SImmetry Sacroiliac Joint Fusion System.

DETAILED DESCRIPTION:
This is a prospective, non-randomized post market study designed to evaluate fusion and pain reduction following the use of the SImmetry System. This study will be conducted at up to 40 sites and 250 total subjects will be enrolled and followed through 24 months. Data will be collected pre-operatively, implant, and at specified follow-up time points through 24 months.

ELIGIBILITY:
Key Inclusion Criteria:

* At least three positive provocative tests for SIJ pain
* Non-operative management of SIJ pain for ≥ 6 months prior to surgery
* At least one positive diagnostic SIJ injection resulting in a ≥ 50% decrease in pain
* VAS back pain score of ≥ 60 mm
* The subject is at least 18 years of age

Key Exclusion Criteria:

* Trauma causing fracture of the sacrum or iliac bones or has had spinal trauma leading to a neurological deficit, or pelvic soft tissue or bony tumors
* Pregnant or is planning on becoming pregnant in the next two years
* Chemical dependency abuse problems as evidenced by a history of abusing drugs which is documented in their past medical history or is elicited from an interview.
* Receiving or seeking worker's compensation, disability remuneration, and/or involved in litigation related to low back or SIJ pain
* History of significant emotional or psychosocial disturbance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Investigator's standard patient population diagnosed with SIJ pain and representing candidates for SIJ fusion.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
SI Joint Fusion | 12 months
  Fusion of the SI joint at 12 and 24 months, defined as presence of a continuous segment of solid bridging bone that extends from the sacrum to the ilium. This will be assessed by an independent core laboratory
SI Joint Pain Reduction | 6 Months
  SI joint pain reduction evaluated by use of Visual Analogue Scale (VAS) for back pain for comparison of baseline to 6 months.

SECONDARY OUTCOMES:
SI Joint Pain Reduction | 12 months
  SI joint pain reduction evaluated by use of Visual Analogue Scale (VAS) for back pain for comparison of baseline to all follow-up visits.
Disability | 6 months
  Functional ability as determined by the Oswestry Disability Index
Quality of Life | 6 months
  Quality of life as determined by EQ-5D

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - The CORE Institute, Phoenix, Arizona
  - BASIC Spine, Newport Beach, California
  - Kaiser Permanente, Oakland, California
  - Rocky Mountain Spine Clinic, Lone Tree, Colorado
  - Orthopaedic Clinic of Daytona Beach, Daytona Beach, Florida
  - Central Florida Neurosurgery Institute, Orlando, Florida
  - Flagler Hospital, Saint Augustine, Florida
  - Gainesville Physical Therapy, Gainesville, Georgia
  - DK Orthopaedics, Crown Point, Indiana
  - SBA Medical Center, El Dorado, Kansas
  - Western Michigan University Homer Stryker MD School of Medicine, Kalamazoo, Michigan
  - Tristate Brain and Spine Institute, Alexandria, Minnesota
  - Essentia Health, Duluth, Minnesota
  - Regional Brain and Spine, Cape Girardeau, Missouri
  - Portland Pain and Spine, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Black Hills Orthopedic & Spine Center, Rapid City, South Dakota
  - Azalea Orthopedics, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Bellevue Bone and Joint Physicians, Bellevue, Washington
  - Fourth Corner Neurological Associates, Bellingham, Washington
  - Northwest Orthopaedic Specialists, Spokane, Washington